CLINICAL TRIAL: NCT03278093
Title: The Feasibility and Effect of Ankle Foot Orthoses and Underfoot Vibration on the Postural Stability of People With Inherited Neuropathy
Brief Title: Effect of Orthoses and Underfoot Vibration on Balance in Neuropathy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: St George's, University of London (Other)
Collaborators: University College London Hospitals (Other)
Responsible Party: Sponsor
Other Study IDs: 16.0029
Record Dates: First submitted 2017-09-08; First posted 2017-09-11 (Actual); Last update posted 2019-01-22 (Actual); Status verified 2019-01

CONDITIONS: CMT - Charcot-Marie-Tooth Disease; Peripheral Neuropathy; Hereditary Peripheral Neuropathy; CMT1A
Keywords: Physiotherapy; Physical therapy; Balance; Posturography
MeSH Terms: conditions — Charcot-Marie-Tooth Disease; Peripheral Nervous System Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A cross-sectional study which will look at the effects of AFO's and vibrating insoles on balance performance in people with CMT disease.

DETAILED DESCRIPTION:
Balance impairments and falls are more common in people who have Charcot Marie Tooth disease (CMT) than in people without the condition. CMT is a condition which affects the nerves causing a variety of symptoms including sensation impairments and weakness. The impairments are usually most evident in the feet and hands, but they can progress very slowly moving closer to the trunk. Ankle Foot Orthoses (AFO's) are often prescribed to help with walking and daily function. So far the effects of AFO's on standing balance in people who have CMT have not been looked at. Insoles are also often prescribed to realign foot deformity and reduce pain. Insoles which give a vibratory input have had a positive impact on walking in older people but have not been looked at in balance and in CMT. Insoles which give a vibration feedback to the sole of the foot when worn have been designed. This study will look at whether the use of AFO's and the vibratory insoles have an effect on standing balance in people with CMT or related peripheral neuropathy. Balance measurements will be taken in a single session comparing a variety of postures. Patients will be recruited from neurology outpatient clinics at the National Hospital of Neurology and Neurosurgery.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical or genetically confirmed diagnosis of CMT or related peripheral neuropathy
2. Mixed sensory and motor presentation
3. Over 18 years
4. Able to stand unsupported for five minutes
5. Able to walk for 50m with or without a walking stick or orthotic devices

Exclusion Criteria:

1. Presence of other significant neurological disorders (such as multiple sclerosis, cerebrovascular diseases, epilepsy, movement disorders), or major comorbidities (e.g. vestibular dysfunction, use of medication which may affect balance, cognitive impairment, presence of medical conditions in which exercise training may be detrimental).
2. Presence of peripheral neuropathy caused by a condition other than CMT.
3. Limb surgery during the six months prior to screening (or planned before final assessment).
4. Women of child-bearing age if they are pregnant, planning a pregnancy during their time in the study or in the 12 weeks following giving birth. This is due to the effects of pregnancy on balance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Mobile adults who have CMT with both motor and sensory symptoms.
Sampling Method: Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2017-10-20 (Actual); Primary Completion 2019-02-20 (Estimated); Study Completion 2019-02-20 (Estimated)

PRIMARY OUTCOMES:
Posturography | 30 second caputer in a variety of conditions
  CODA motion movement analysis for postural sway Measures will be taken in all conditions with feet together and feet apart. Both conditions will also be looked at with eyes open and eyes closed.
force measures | 30 second caputer in a variety of conditions
  AMTI forceplate for centre of pressure . Measures will be taken in all conditions with feet together and feet apart. Both conditions will also be looked at with eyes open and eyes closed.

CONTACTS AND LOCATIONS:
Overall Officials: Gita Ramdharry, Principal Investigator — Senior Physiotherapist
Locations (1):
- National Hopsital of Neurology and Neurosurgery, London, United Kingdom